CLINICAL TRIAL: NCT00531869
Title: A Study of End-User Preferences for and Use of POU Safe Water Technologies in Kenya
Brief Title: Safe Water Techniques in Kenya
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, Berkeley (Other)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Dr. David I Levine, UC Berkeley CEGA
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CPHS Protocol #2007-7-27
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Last update posted 2008-08-04 (Estimated); Status verified 2008-07

CONDITIONS: Consumer Willingness to Pay for POU Products; Consumer Preferences and Use of POU Products
Keywords: safewater; randomized
MeSH Terms: conditions — Consumer Behavior

INTERVENTIONS:
Behavioral: biases towards products

SUMMARY:
Consumer preferences for POU technologies vary across consumers and products, and largely determine their adoption and subsequent usage. This is a marketing study that asks which products consumers prefer and why, and what is their willingness to pay, as understanding this is crucial to attain their widespread adoption and usage.

DETAILED DESCRIPTION:
Visit 400 households and distribute 1 of 3 different POU technologies on randomized basis for a two-month trial. Cycle each household through trials with all 3 technologies in random order such that at the end of 6 months all households have experienced 2-month trials with each technology.

ELIGIBILITY:
Inclusion Criteria:

* At least partial reliance on turbid water supply

Exclusion Criteria:

* At least partial reliance on turbid water supply

Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 2008-05; Primary Completion 2010-05 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Consumer preferences and use of POU products

SECONDARY OUTCOMES:
Consumer willingness to pay for POU products

CONTACTS AND LOCATIONS:
Overall Officials: David Levine, PhD Econ, Principal Investigator — UC Berkeley
Locations (1):
- Care Kenya, Kisumu, Kenya